CLINICAL TRIAL: NCT01294280
Title: Participation in the Lung Adjuvant Cisplatin Evaluation Biological Program (LACE-BIO). A Study of Prognostic and Predictive Markers in Early Stage Non-Small Cell Lung Cancer
Brief Title: Biomarkers in Predicting Response in Patients With Early-Stage Non-Small Cell Lung Cancer Previously Treated With Adjuvant Chemotherapy
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150802; CDR0000600208 (Registry Identifier: NCI Physician Data Query); U10CA031946 (NIH); NCI-2009-00454 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer
Keywords: Stage I Non-Small Cell Lung Cancer; Stage II Non-Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (IHC): Previously collected tissue samples are analyzed by IHC.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies prognostic and predictive markers in patients with early stage non-small cell lung cancer receiving chemotherapy. Prognostic markers are patient or tumor factors that predict patient survival independent of treatment. Predictive markers are factors that may influence and predict the outcome of treatment in terms of either response or survival benefit. Collecting and storing samples of tissue from patients with cancer to study in the laboratory may help doctors learn more about cancer and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate potential prognostic and predictive markers in patients receiving adjuvant chemotherapy for early stage non-small cell lung cancer (NSCLC).

II. To perform cross-validation analyses for the predictive value of cyclin-dependent kinase inhibitor 1B (p27), excision repair cross-complementation group 1 (ERCC1), beta-tubulin and B-cell lymphoma 2 (BCL2)-associated X protein (BAX).

III. To perform cross-validation analyses for the prognostic value of mucin and breast cancer (BRCA)1 expression.

IV. To perform a pooled analysis for the prognostic impact of p53 protein expression by immunohistochemistry (IHC), tumor protein p53 (p53) mutation, ras mutation and epidermal growth factor receptor (EGFR) mutation, and Fas cell surface death receptor (Fas)/Fas ligand (FasL) expression by IHC.

V. Validation of the 15-gene prognostic and predictive messenger ribonucleic acid (mRNA) signature on Lung Adjuvant Cisplatin Evaluation (LACE)-Bio formalin-fixed paraffin-embedded (FFPE) tumor samples.

VI. Exploratory evaluation of the prognostic and predictive values of known potential oncogenic mutations using LACE-Bio FFPE.

VII. Exploratory evaluation of the prognostic and predictive values of gene copy variation using LACE-Bio FFPE tumor samples.

VIII. Exploratory identification and evaluation of prognostic and predictive value of novel genomic aberrations discovered by Next Generation Sequencing on LACE-Bio tumor samples.

OUTLINE:

Previously collected tissue samples are analyzed by IHC.

ELIGIBILITY:
Inclusion Criteria:

* Registration to CALGB9633 for this study
* Institutional Review Board (IRB) review and approval at the institution where the laboratory work will be performed is required
* Informed consent:

  * The subject population to be studied in this protocol includes patients selected from CALGB 9633 for whom an available specimen is present at the Alliance Ohio State University (OSU); all such patients have signed a written informed consent document meeting all federal, state, and institutional guidelines as part of entry into that trial
  * Only cases with adequate tumor formalin FFPE material without depleting the available clinical block(s) are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients registered to Cancer and Leukemia Group B (CALGB) 9633
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2016-02-02 (Actual); Study Completion 2016-02-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 3 years

SECONDARY OUTCOMES:
Disease-free survival | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Graziano, MD, Study Chair — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States